CLINICAL TRIAL: NCT03305913
Title: Regorafenib in Combination With TAS-102 in Subjects With Metastatic Colorectal Cancer Who Have Progressed After Standard Therapy: A Multicenter Phase I Study
Brief Title: Regorafenib in Combination With TAS-102 in Subjects With Metastatic Colorectal Cancer Who Have Progressed After Standard Therapy
Acronym: REMETY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Institut für Klinisch-Onkologische Forschung (IKF) am Krankenhaus Nordwest GmbH (Unknown); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0116-ASG; 2016-001968-11 (EudraCT Number)
Record Dates: First submitted 2017-08-16; First posted 2017-10-10 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Pretreated Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: interventions — trifluridine tipiracil drug combination; regorafenib

STUDY DESIGN:
Intervention Model Description: According to the standard 3+3 dose finding strategy, a safety assessment will be performed after the test of each dose level (patient cohorts of n=3) and the frequency of DLTs determined. Based on the results the dose for the consecutive patient cohort will either be escalated (0/3 DLTs), repeated (1/3 DLTs) or deescalated (>1/3 DLTs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Experimental): TAS-102 25 mg/m2 BID (days 1-5 and 8-12) Regorafenib 120 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib
- Dose Level 2 (Experimental): TAS-102 35 mg/m2 BID (days 1-5 and 8-12), Regorafenib 120 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib
- Dose Level 3 (Experimental): TAS-102 35 mg/m2 BID, (days 1-5 and 8-12) Regorafenib 160 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib
- Dose Level -1a (Experimental): TAS-102 25 mg/m2 BID, (days 1-5 and 8-12) Regorafenib 80 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib
- Dose Level -1b (Experimental): TAS-102 35 mg/m2 BID, (days 1-5 and 8-12) Regorafenib 80 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib
- Dose Level -2a (Experimental): TAS-102 30 mg/m2 BID (or 35 mg/m2 a.m. and 25 mg/m2 p.m.), (days 1-5 and 8-12) Regorafenib 120 mg daily (3 weeks on, 1 week off)
  Interventions: Drug: TAS 102; Drug: Regorafenib

INTERVENTIONS:
Drug: TAS 102 — TAS-102 tablet
  Other Names: Lonsurf
Drug: Regorafenib — Regorafenib tablet
  Other Names: Stivarga

SUMMARY:
0116-ASG REMETY is a multicenter, open-label, non-randomized, dose-escalation Phase I study evaluating the safety and anti-tumor activity of TAS-102 administered in combination with Regorafenib in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
The primary objective is to determine safety, feasibility and the recommended phase II dose (RP2D) of a combination treatment consisting of TAS-102 and Regorafenib in subjects with mCRC who have progressed after standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Histological or cytological documentation of adenocarcinoma of the colorectal region (CRC)
4. Metastatic disease not amenable to surgical resection with curative intent
5. Study treatment must constitute 3rd-line treatment for metastatic disease. Prior treatment lines must encompass at least one fluoropyrimidine-based chemotherapy, an anti-VEGF and, in case of RAS wildtype tumors, an anti-EGFR treatment.
6. Patients treated with oxaliplatin in an adjuvant setting need to have progressed during or within 6 months of completion of adjuvant therapy to be counted as prior treatment line. Note: Neoadjuvant, perioperative or adjuvant regimens with progression more than 6 months after completion are not considered as prior treatment line for metastatic disease.
7. Measurable disease, defined as at least one unidimensional measurable lesion on a CT scan as defined by RECIST 1.1
8. Eastern Cooperative Oncology Group (ECOG) performance status <2 and life expectancy of at least 3 months
9. Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days prior to study treatment initiation:

   * Absolute neutrophil count (ANC) ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Serum creatinine ≤1.5 x upper limit of normal (ULN)
   * Glomerular filtration rate (GFR) ≥30 mL/min/1.73m2
   * AST and ALT ≤2.5 x ULN (≤5.0 × ULN for patients with liver involvement of their cancer)
   * Bilirubin ≤1.5 X ULN
   * Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN with liver involvement of their cancer)
   * Amylase and lipase ≤1.5 x ULN
   * Spot urine must not show 1+ or more protein in urine or the patient will require a repeat urine analysis. If repeated urinalysis shows 1+ protein or more, a 24-hour urine collection will be required and must show total protein excretion <1000 mg/24 hours
   * INR/PTT ≤1.5 x ULN (Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.)
10. Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation and up to 6 months following completion of therapy. Females of childbearing potential who are sexually active with a non-sterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for 6 months after the final dose of investigational product.
11. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a pregnancy test performed at a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
12. In the assessment of the investigator, patient is able to comply with study requirements.
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Prior treatment with Regorafenib, or any other tyrosine kinase inhibitor for the treatment of malignancy
2. Prior treatment with TAS-102
3. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to study inclusion EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (Non invasive tumor), Tis (Carcinoma in situ) and T1 (Tumor invades lamina propria)].
4. Known history of/or concomitant malignancy other than mCRC likely to affect life expectancy in the judgment of the investigator
5. History of Gilbert's syndrome
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days and last chemotherapy <21 days prior to first dose of treatment
7. Radiotherapy within 4 weeks prior to first dose of treatment
8. Active cardiac disease including any of the following:

   * Congestive heart failure (New York Heart Association NYHA) ≥Class 2
   * Unstable angina (angina symptoms at rest), new-onset angina (within the last 3 months).
   * Myocardial infarction less than 6 months before start of Day 1 of treatment.
   * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
   * Uncontrolled hypertension. (Systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
9. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before start of treatment
10. Known history of human immunodeficiency virus (HIV) infection
11. Chronic hepatitis B or C infection (If hepatitis status can not be obtained from medical records re-testing is required.)
12. Patients with seizure disorder requiring medication
13. Symptomatic metastatic brain or meningeal tumors unless the patient is >6 months from definitive therapy, has a negative imaging study within 4 weeks prior to treatment initiation, and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable, provided that the dose is stable for one month prior to and following screening radiographic studies).
14. History of organ allograft
15. Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ Grade 3 (CTCAE v. 4.0) within 4 weeks prior to the start of study treatment.
16. Non-healing wound, ulcer or bone fracture
17. Renal failure requiring hemo- or peritoneal dialysis
18. Dehydration according to CTCAE v. 4.03 Grade >1
19. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
20. Known hypersensitivity to any of the study drugs, study drug classes, or any constituent of the products
21. Known dihydropyrimidine dehydrogenase (DPD) deficiency or treatment with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine within 4 weeks prior to the start of study treatment.
22. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
23. Inability to swallow oral medications
24. Any malabsorption condition
25. Unresolved toxicity higher than Grade 1 CTCAE v. 4.03 attributed to any prior therapy/procedure excluding alopecia, anemia and oxaliplatin-induced neurotoxicity (which must be ≤Grade 2) or ongoing infection >Grade 2.
26. Patients unable or unwilling to discontinue (and substitute if necessary) use of prohibited drugs for at least 2 weeks prior to Day 1 of treatment initiation.
27. Female subjects who are pregnant, breast-feeding or intent to become pregnant
28. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
29. Participation in another clinical study with an investigational product during the last 30 days before inclusion
30. Previous enrollment in the present study (does not include screening failure).
31. Involvement in the planning and/or conduct of the study (applies to Bayer staff and/or staff of sponsor and/or staff of the CRO and study site)
32. Patient who might be interconnected with or dependent on the sponsor, site or the investigator Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 months
  Maximum Tolerated Dose (MTD) will be determined by recording dose limiting toxicities (DLT) occurring during the first 2 treatment cycles of each patient in each tested dose level. DLT will be identified by observing frequency and severity of specific adverse events.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to RECIST 1.1 criteria | approx. 12 months
  ORR is defined as the proportion of ALL Treated Subjects whose best overall response (BOR) from baseline is either a CR or PR per RECIST 1.1 criteria. BOR is determined by the best response designation recorded between the date of subject enrollment and the date of objectively documented progression. For subjects without documented progression, all available response designations will contribute to the BOR determination.
  ORR will be evaluated by reporting absolute and relative frequencies.
Progression-free survival (PFS) | approx. 12 months
  Progression free survival will be calculated from the date of subject enrollment until the date of confirmed PD or death from any cause. If no event is observed (e.g. lost to follow-up) PFS is censored at the time of last tumor assessment.
Overall survival (OS) | approx. 12 months
  Overall Survival will be calculated from the date of subject enrollment until the date of death from any cause. If no event is observed (e.g. lost to follow-up) OS is censored at the day of last subject contact.
Incidence of Treatment-Emergent Adverse Events | approx. 12 months
  Incidence of AEs, SAEs, Treatment Emergent Adverse Events according to CTC 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Markus Möhler, Prof. Dr., Principal Investigator — Universitätsmedizin Mainz, I.Medizinische Klinik und Poliklinik, Langenbeckstraße 1, 55131 Mainz
Locations (1):
- Universitätsmedizin Mainz, I.Medizinische Klinik und Poliklinik, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moehler M, Michel M, Stein A, Trojan J, Marquardt J, Tintelnot J, Waidmann O, Weinmann A, Woerns MA, Schroeder H, Maenz M, Foerster F. A Phase I dose-escalation study of third-line regorafenib with trifluridine/tipiracil in metastatic colorectal cancer. Future Oncol. 2021 Sep;17(25):3309-3319. doi: 10.2217/fon-2021-0278. Epub 2021 May 17. PMID 33993741